CLINICAL TRIAL: NCT06558955
Title: Technology-enabled Anticipatory Guidance and Peer Support in Empowering Parents to Prevent Early Childhood Caries: A Randomized Controlled Trial
Brief Title: Technology-enabled Anticipatory Guidance and Peer Support in Empowering Parents to Prevent Early Childhood Caries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Gao Xiaoli, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DSRB 2024/00244; PHRGOC23jul-0011 (Other Grant/Funding Number: National Medical Research Council, Singapore)
Record Dates: First submitted 2024-07-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries; Dental Caries in Children; Diet Habit
Keywords: Anticipatory Guidance; Peer Support; Oral Health; Technology; Dental Caries
MeSH Terms: conditions — Dental Caries; Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-enabled anticipatory guidance and peer support (Experimental): Participants (mothers) will join online parent empowerment sessions for about 4 times (around 3, 6, 12, and 18 months of child's age, around 45 - 60 minutes each), and receive additional information and push notifications via a mobile phone app.
  Interventions: Behavioral: Technology-enabled anticipatory guidance and peer support
- Conventional oral health education (Active Comparator): Participants (mothers) will receive child oral health information for about 4 times (around 3, 6, 12, and 18 months of child's age).
  Interventions: Behavioral: Conventional health education

INTERVENTIONS:
Behavioral: Technology-enabled anticipatory guidance and peer support — The intervention includes 4 online sessions led by an oral health therapist (OHT) or dentist, as well as push notifications and information delivered to participants via a mobile/web app.
  Arms: Technology-enabled anticipatory guidance and peer support
Behavioral: Conventional health education — Participants on this arm will receive conventional child oral health education materials at 4 time points.
  Arms: Conventional oral health education

SUMMARY:
Early Childhood Caries (ECC) is a significant clinical and public health challenge that the world and the Singapore population are facing. This study seeks to test the effectiveness of technology-enabled anticipatory guidance and peer support in empowering parents to establish proper childcare practices and prevent ECC.

DETAILED DESCRIPTION:
The study design is a two-arm, parallel group, assessor-blinded, randomised controlled trial. The hypothesis is that technology-enabled anticipatory guidance and peer support is more effective than conventional oral health education in enhancing parental efficacy, establishing proper childcare practices (dietary, feeding and toothbrushing), and preventing ECC. Up to 600 mother-child dyads will be recruited and randomly assigned to receive conventional oral health education (control), and technology-enabled anticipatory guidance and peer support (intervention), respectively. For the intervention arm, anticipatory guidance and peer support will be delivered through 4 unique online sessions for mothers, when each child turns 3, 6, 12, and 18 months, to match the developmental milestones and parental needs for childcare support. Outcomes will be assessed through a questionnaire and food diary (at 12, 24 and 36 months of child's age) and a dental examination for the child (at 24 and 36 months of age).

The effectiveness of the intervention will be evaluated using psychological outcomes (parental efficacy), behavioral outcomes (dietary, feeding and oral hygiene practices), and clinical outcomes (oral hygiene and ECC), and quality of life outcomes. Process evaluation and cost-effectiveness analysis will be included. Data will be analyzed on an intention-to-treat basis, including with the last observation carried forward method. Descriptive statistics on socio-demographic backgrounds, parental efficacy, childcare practices, child's oral health status, and oral health related quality of life will be reported. Chi-square test and two-sample t-test, or their non-parametric equivalents, will be used as appropriate to compare proportions and means between the control and intervention groups. Effect sizes and number needed to be treated will be presented to provide an estimate of the number of parents needed to be intervened in order to avoid one child with new dental caries. Multivariable analyses will be performed to evaluate the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Mother is currently expecting or has an infant below 3 months of age
* Biological mother of the child
* Mother with internet access and a mobile device
* Mother can communicate in English
* Mother aged 21 years and above

Exclusion Criteria:

* Child with disqualifying medical condition (e.g., tube feeding, severe neuromuscular disability) that would limit oral dietary intake, at-home oral hygiene practices, or receipt of dental examinations
* Child with serious congenital syndrome that is expected to adversely affect the development of primary teeth
* Family plans to emigrate within 3 years

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of early childhood caries | 24 and 36 months of age for children
  Number of new surfaces with coronal caries

SECONDARY OUTCOMES:
Toothbrushing behaviours | 12, 24 and 36 months of age for children
  Using a questionnaire, toothbrushing behaviours will be categorised as:
  1. Favourable (frequency of brushing >=2times/day)
  2. Unfavourable (frequency of brushing <2times/day)
Dietary and feeding practices (favourable/unfavourable) | 12, 24 and 36 months of age for children
  Self-reported frequency of snack, sweet/dessert and sugary drink intake
Dental Utilisation | 12, 24 and 36 months of age for children
  Self-reported frequency of dental visits
Dental Costs | 12, 24 and 36 months of age for children
  Sum of direct costs from dental treatment and indirect costs due to time taken off work by parents to attend dental visits, and loss of productivity. Costs will be captured in Singapore dollars (SGD).
Parental efficacy in managing oral health of child | 12, 24 and 36 months of age for children
  Measured using the self-efficacy scale for maternal oral care (SESMO). Response options ("Yes" and "No"). A score of 1 is given for an answer with higher self-efficacy and 0 for lower self-efficacy. Minimum score is 0 and maximum score is 16 for the 16 questions. Higher scores indicate better outcomes.
Plaque score | 24 and 36 months of age for children
  Plaque score based on the index recommended by Ramjford and modified for primary dentition. The plaque score is coded as following: 2 = visible plaque without use of probe, 1 = no visible plaque but a probe skimmed over the tooth surface reveals plaque, 0 = no plaque. Scoring is done at three sites (interproximal, buccal and palatal/lingual) on the index teeth (#54, #61, #64, #74, #81, #84).
Breastfeeding rate | 12 and 24 months of age for children
  Duration of breastfeeding (in months)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Gao, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao X, Tan SHX, Hong CHL, Chong MFF, Wong ML, Ng YPM, Koh GCH, Foong PS, Pramanick A, Eu OC, Gallagher JE, Amin Z. Technology-enabled anticipatory guidance and peer support in empowering parents to prevent early childhood caries: a randomized controlled trial. BMC Oral Health. 2024 Dec 4;24(1):1470. doi: 10.1186/s12903-024-05204-7. PMID 39633367